CLINICAL TRIAL: NCT06290622
Title: PD-1, LAG-3 and TIM-3 Checkpoint Blockade in DLBCL Post Chimeric Antigen Receptor T-cEll Therapy fAilUre (PLATEAU Study)
Brief Title: PD-1, LAG-3 and TIM-3 Checkpoint Blockade in DLBCL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Investigator request to no longer pursue this study. Lack of support from drug company. This trial never opened. Withdrew IND.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mayur Narkhede, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB300012414 (UAB23136)
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Lymphoma, B-Cell; Lymphoma, Follicular
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Level Assignments (Experimental): Dose Level 1 Retifanlimab 375mg INCAGN02385 250mg INCAGN02390 200mg
  Dose Level 2 Retifanlimab 500mg INCAGN02385 250mg INCAGN02390 200mg
  Dose Level 3 Retifanlimab 750mg INCAGN02385 250mg INCAGN02390 200mg
  Interventions: Drug: Retifanlimab, INCAGN02385, INCAGN02390

INTERVENTIONS:
Drug: Retifanlimab, INCAGN02385, INCAGN02390 — Treatment:
  Retifanlimab -infused over 60 minutes for C1D1 followed by a 60-minute observation period. If no infusion related reactions are observed infusion may be reduced to 30 minutes and no further observation period is needed for future cycles. If there is a reaction continue with 60 minute infusion and observation period for following cycle. Retifanlimab should always be administered first.
  INCAGN02385 and INCAGN02390 -individually administered over 30 minutes one after another. For first infusions of retifanlimab, INCAGN02385 and INCAGN02390, a 4 hour observation period is necessary after completion of all infusion. If no infusion related reactions are observed, for subsequent infusions no further observation period is needed for future cycles.

SUMMARY:
This study is investigating the optimal dose and the advantage in combining investigational immunotherapy drugs known as Retifanlimab, INCAGN02385 and INCAGN02390 to improve the responses to CAR T-cell therapy. Additionally, the study will investigate that triple checkpoint blockade of PD-1, TIM-3 and LAG-3 molecules will overcome CAR T-cell therapy resistance in patients with suboptimal responses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have received CAR T-cell therapy within 120 days as per the United States Food and Drug Agency (USFDA) approved indications for

   * Diffuse large B-cell lymphoma (DLBCL),
   * Primary mediastinal large B-cell lymphoma (PMBCL),
   * High grade B-cell lymphoma,
   * DLBCL arising from indolent lymphoma.
   * Follicular Lymphoma Grade 3B.

   Who receieved a CD19 directed CAR T-cell therapy product of any of the following
   * Axicabtagene Ciloleucel (Axi-cel)
   * Tisagenlecleucel (Tisa-cel)
   * Lisocabtagene Ciloleucel (Liso-cel)
2. Patients with persistent or refractory disease with a Deauville score of 4 or 5 as per Lugano Criteria or early relapse within 90 days after CAR T-cell therapy.
3. Adequate organ function as defined below unless attributed to disease involvement.

   1. liver function (bilirubin < 2mg/dL, AST and/or ALT <3 x ULN)
   2. kidney function (crcl > 30ml/min using Cockroft-Gault, based on actual weight).
   3. ANC ≥ 1,000/µL, Hgb > 8, Platelet Count ≥ 50,000/ µL. Transfusions allowed. Growth factor support allowed.
   4. TnT or TnI < 2 × Institutional ULN. Participants with TnT or TnI levels between > 1 to 2 × ULN will be permitted if repeat levels within 24 hours are ≤ 1 × ULN.
4. Patients with HIV can be included if they are on appropriate antiretroviral therapy, a CD4+ T-cell counts ≥ 300 cells/µL and no detectable viral load.
5. Age ≥ 18 years of age.
6. Eastern Cooperative Group performance (ECOG) status of 0 to 2.
7. A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial.
8. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 months after infusion of study drug.
9. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.
10. Willing and able to participate in all required evaluations and procedures in this study protocol including receiving intravenous administration of investigational product and being admitted, when required, for at least 24 hours during investigational product administration.

Exclusion Criteria:

1. Patients who experienced Grade 3 or higher Cytokine release syndrome (CRS) or Immune cell associated neurotoxicity syndrome (ICANS) with CAR T-cell therapy as per ASTCT criteria.
2. Patients with ongoing CRS or ICANS.
3. Patients who experienced hemophagocytic lymphohistiocytosis (HLH) due to CAR T- cell therapy.
4. Prior allogeneic stem cell transplant within 6 months. The patient should not have any active Graft vs. Host disease (GVH) or should be on immune suppressive agents.
5. Prior treatment with PD-(L)1, TIM-3 or LAG-3 blocking therapy.
6. Any active, concurrent, significant illness or disease (other underlying lymphoma) or clinically significant findings including psychiatric and behavioral problems, medical history and/or physical examination findings that would preclude the patient from participation in the study such as:

   * active infection requiring systemic therapy ≤14 days before the first dose of study drug
   * unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association [NYHA] II, III, IV;), myocardial infarction ≤6 months prior to first study drug, uncontrolled cardiac arrhythmia e.g., atrial fibrillation/flutter, cerebrovascular accidents ≤6 months before first dose of study drug
   * Significant (as defined by study doctor) pulmonary disease or disorder, including interstitial lung disease or history of interstitial lung disease, or active, noninfectious pneumonitis.
   * Severe autoimmune disorder with evidence of significant organ damage from autoimmune disorder as defined by study physician.
   * any severe or uncontrolled other disease or condition which might increase the risk associated with study participation.
   * History of myocarditis as defined by a cardiologist requiring immunosuppressive therapies.
   * Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath) and not related to underlying lymphoma.
7. Vaccination with live, attenuated vaccines within 28 days prior to the first dose of study medication.
8. Patients who develop COVID-19 (SARS-CoV2) infection at any time during screening, should not be enrolled until a negative PCR is confirmed and all clinical symptoms (as applicable) have resolved.
9. Receiving systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents). The use of inhaled corticosteroids is permitted.
10. Corticosteroids ≥ 10 mg of prednisone within 7 days of first dose of study drug.

    Notes:
    1. Physiologic corticosteroid replacement therapy at doses > 10 mg/day of prednisone or equivalent for adrenal or pituitary insufficiency and in the absence of active autoimmune disease is permitted.
    2. Participants with a condition (eg, asthma or COPD) that requires intermittent use of bronchodilators, inhaled steroids, or local steroid injections may participate.
    3. Participants using topical, ocular, intra-articular, or intranasal steroids (with minimal systemic absorption) may participate.
    4. Brief courses of corticosteroids for prophylaxis (e.g., contrast dye allergy) or study treatment-related standard premedication are permitted.
11. Has known active HBV or HCV infection, or risk of reactivation of HBV or HCV, defined as follows (testing must be performed to determine eligibility):

    - Active HBV infection is defined by positive HBsAg and positive total anti-HBc results.

    Note: When HBsAg is negative AND HBcAb and/or HBsAb is positive, HBV-DNA should be measured. When HBV-DNA is negative, this participant could be enrolled with close monitoring of HBV activities.

    - Active HCV is defined as a positive HCV antibody result and quantitative HCV-RNA results greater than the lower limits of detection of the assay.

    Note: Participants positive for HCV antibody will be eligible if they are negative for HCV-RNA. Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable.
12. Patients with prior solid organ transplant
13. Breastfeeding or pregnant
14. Any other malignancy known to be active, with the exception of

    * Cervical carcinoma of Stage 1B or less
    * Non-invasive basal cell or squamous cell skin carcinoma
    * Non-invasive, superficial bladder cancer
    * Prostate cancer with a current PSA level < 0.1 ng/mL
    * Any curable or localized cancer with a CR of > 2 years' duration.
15. Known allergy or hypersensitivity to any component of either retifanlimab, INCAGN02385, or INCAGN02390 study drug formulation (including excipients and additives). Patients with known hypersensitivity to another monoclonal antibody that cannot be controlled with standard measures such as antihistamines and/or corticosteroids will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Identify the optimal biological dose (OBD) for Retifanlimab in combination with INCAGN02385 and INCAGN02390 in relapsed/refractory DLBCL. | 12 and 24 months
  To find the dose at which efficacy and toxicity are balanced to obtain a desirable dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mayur Narkhede, Principal Investigator — University of Alabama at Birmingham